CLINICAL TRIAL: NCT01509599
Title: Preventing Venous Leg Ulcers With Cryotherapy: A Randomized Clinical Trial
Brief Title: Cooling Lower Leg Skin to Prevent Venous Leg Ulcers in Patients With Poor Vein Circulation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Teresa Kelechi, Associate Professor and Department Chair, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00008711; 1R01NR012237-01A1 (NIH)
Record Dates: First submitted 2011-08-19; First posted 2012-01-13 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Venous Disease; Venous Vascular Diseases and Syndromes; Venous Insufficiency; Venous Ulcers
Keywords: Venous disease; Venous disorders; Venous insufficiency; Venous ulcers; Cryotherapy
MeSH Terms: conditions — Syndrome; Venous Insufficiency; Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryotherapy (Experimental): Cryotherapy is delivered via a cooling "gel" wrap applied to the affected lower leg using a dosing regimen, starting with daily cooling in month one to PRN in the last 3 months over the 9 month study.
  Interventions: Procedure: Cryotherapy: Cooling gel wrap
- Usual care (Sham Comparator): The "sham" wrap, filled with cotton, is applied to the affected lower leg using a dosing regimen, starting with daily application in month one to PRN in the last 3 months over the 9 month study.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Cryotherapy: Cooling gel wrap — Patients will wear compression stockings (provided), elevate legs on an elevator pillow (provided) and apply the sham cyrotherapy: cooling gel wrap during the home-based intervention
  Other Names: Cooling cuff, cool cuff
  Arms: Cryotherapy
Procedure: Usual care — Patients will wear compression stockings (provided), elevate legs on an elevator pillow (provided) and apply the sham cyrotherapy wrap (sham) during the home-based intervention
  Other Names: Standard of care; Guideline guided care
  Arms: Usual care

SUMMARY:
Leg vein circulation problems can damage the skin of the lower legs, especially around the ankles, by making it discolored, hard, itchy, red, and swollen. Ulcers often develop. Inflammation is often present in the damaged skin. This study will test whether using a special low compression, cooling, boot-like gel wrap placed around the damaged skin of the lower legs will improve the skin circulation and prevent leg ulcers. The study hypothesis is: A cryotherapy, low-compression cooling gel wrap (CW) plus usual care (UC) (leg elevation, compression stockings) intervention compared to a low compression non-cryotherapy "sham" wrap (NW) plus UC will reduce tissue blood flow (perfusion units) and decrease the incidence of venous leg ulcers (VLUs) during the 9-month study period in individuals with Stage 4 and 5 venous insufficiency.

DETAILED DESCRIPTION:
This new trial will assess the efficacy of this home-based cryotherapy intervention by adding sequenced tapered cooling after a 30-day intense cooling period. The goal is to reduce skin blood flow of chronically inflamed skin, decrease the incidence of venous leg ulcers and pain, and improve quality of life. A myriad of surgical, pharmacologic, and non-pharmacologic therapies such as compression bandages are often tried, many with limited success. More than 70% of patients with venous disorders such as insufficiency develop edema, skin damage, and ulcers. Ulcer prevention is warranted because of the significant socioeconomic implications in terms of lost workdays and wages, decreased productivity and increased health care costs. Clinicians focus on the multiple treatment approaches, often without consideration of how patients can contribute to their own self-care. Our 9-month intervention is based on principles of heat transfer and cryotherapy theories involving microcirculation. With input from a cryotherapy expert and participants who completed the R21 pilot, the investigators propose a sequenced intervention strategy, where cooling will be dosed daily for 30 minutes for the first month, and then decreased to twice weekly dosing in months 2-3, once weekly in months 4-6, then PRN in months 7-9. The investigators will measure blood flow, skin temperature, pain, quality of life, and the incidence of leg ulcers after months 1, 3, 6 and 9. Eligible participants will be randomized to treatment (low compression cooling wrap) or usual care (low compression non-cooling "sham" wrap). Participants in both groups will receive all study related materials including standardized instruction, skin thermometer, specially designed low compression wraps, leg elevator pillow, and compression stockings, and during an in-depth orientation session. The investigators hypothesize that cryotherapy will enhance the largely ineffective non-pharmacologic self-care usual care model, that is, telling patients to wear compression stockings, elevate the legs, and get more exercise. These strategies are generally inadequate in achieving sustained change. Among our research methods the investigators include rigorous process, impact and outcome monitoring. In an era of expectation for technological and pharmaceutical "fixes", this self-care strategy, if efficacious, could be an economical way to decrease morbidity and pain for thousands of patients, frequently viewed as non-responsive to self care. Prevention of ulcers is also a major potential source of saved medical dollars. This trial is significant due to the burden of venous disorders, the complex physical characteristics of the population including excessive obesity and co-morbidity and the need to reach patients with a feasible, motivational, and supportive strategy to promote self-care. The objective is to establish a new practice standard for prevention.

ELIGIBILITY:
Inclusion Criteria:

* aged 21 years or older
* CEAP Classification: Stage C4 (skin damage) and 5 (healed VLU) - leg ulcer healed within past month with intact epithelium
* history of healed VLU within past 2 years
* ankle brachial index (ABI) 0.80 - 1.3 mmHG, absence of peripheral arterial disease
* intact skin sensation
* intact thermal sensation
* agreement to ear compression during waking hours
* phone, email or mail accessible
* willingness to make 5 study visits including baseline
* able to understand protocol by passing test after watching DVD standardized instructions for low literacy
* able to perform required protocol activities
* ability to speak English

Exclusion Criteria:

* diagnosed arterial disease or ABI <0.80 or >1.3 mm Hg (blood flow to the skin is reduced in arterial disease and cooling could cause tissue ischemia)
* surgical procedures on leg in past 1 year (can affect venous circulation/cause edema)
* open leg/foot ulcers
* recent leg infection within past month (increased inflammation)
* impaired cognitive status (cannot perform procedures)
* chronic inflammatory and vascular conditions where blood flow of the skin may be impacted such as Lupus erythematosus, lymphedema, Raynaud's, rheumatoid arthritis, scleroderma, end stage renal disease, chronic obstructive pulmonary disease, chronic regional pain syndrome, multiple sclerosis, hypersensitivity to cold, or patients on chemotherapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Skin blood flow | Skin blood flow will be measured for change at five visits: baseline (visit 1), month 1 (visit 2), month 3 (visit 3), month 6 (visit 4) and 9 (visit 5)
Incidence of venous leg ulcers that develop during the study | Time point will be assessed at months 1, 3, 6 and 9. If an ulcer develops, participants will be followed weekly, for the duration of the ulcer treatment, up to the end of the study at 9 months.
  In the event that a venous leg ulcers develops, the volunteer will notify the study personnel within 24 hours. The volunteer will be instructed to return to the primary care/wound care provider for treatment. Study personnel will contact the volunteer each week to assess progress. If the leg ulcers heals during the time enrolled in the study, the volunteer will continue with the intervention.

SECONDARY OUTCOMES:
Quality of life | During the five measurement points, baseline and then after months, 1, 3, 6, and 9
Pain | Measured at baseline, then after months 1, 3, 6, and 9
Skin temperature | Will be measured daily by the subject and then by student personnel at baseline, then after months 1, 3, 6, and 9

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Data may be requested via the PI and is available through REDCap.

REFERENCES:
- [Background] Kelechi TJ, Johnson JJ, Yates S. Chronic venous disease and venous leg ulcers: An evidence-based update. J Vasc Nurs. 2015 Jun;33(2):36-46. doi: 10.1016/j.jvn.2015.01.003. PMID 26025146
- [Result] Kelechi TJ, Madisetti M, Mueller M, Dooley M, Prentice M. Self-monitoring of lower leg skin temperature: accuracy of self-reported data and adherence to a cooling protocol for the prevention of venous leg ulcers. Patient Prefer Adherence. 2015 Dec 15;9:1751-61. doi: 10.2147/PPA.S91992. eCollection 2015. PMID 26719678
- [Result] Kelechi TJ, Mueller M, King DE, Madisetti M, Prentice M. Impact of daily cooling treatment on skin inflammation in patients with chronic venous disease. J Tissue Viability. 2015 May;24(2):71-9. doi: 10.1016/j.jtv.2015.01.006. Epub 2015 Feb 7. PMID 25703058
- [Result] Kelechi TJ, Mueller M, Dooley M. Sex differences in symptom severity and clusters in patients with stage C4 and stage C5 chronic venous disease. Eur J Cardiovasc Nurs. 2017 Jan;16(1):28-36. doi: 10.1177/1474515116634526. Epub 2016 Jul 7. PMID 26888961
- [Derived] Monsen KA, Kelechi TJ, McRae ME, Mathiason MA, Martin KS. Nursing Theory, Terminology, and Big Data: Data-Driven Discovery of Novel Patterns in Archival Randomized Clinical Trial Data. Nurs Res. 2018 Mar/Apr;67(2):122-132. doi: 10.1097/NNR.0000000000000269. PMID 29489633